CLINICAL TRIAL: NCT01552356
Title: Pharmacokinetic-Driven Individualization of Pazopanib Therapy in Patients With Solid Tumors: A Phase I Study
Brief Title: Pazopanib Hydrochloride in Treating Patients With Advanced or Refractory Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00690; NCI-2012-00690 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MC1112; CDR0000727235; MC1112; MC1112 (Other: Mayo Clinic in Rochester); 9076 (Other: CTEP); P30CA015083 (NIH); U01CA069912 (NIH); UM1CA186686 (NIH); NCT02706366 (obsolete NCT alias)
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Solid Neoplasm
MeSH Terms: interventions — pazopanib

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Course length can be extended to 56 days at the discretion of the treating physician after 12 courses (1 year) of treatment on study.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pazopanib Hydrochloride; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW 786034B; GW-786034B; GW786034B; Pazopater; Votrient
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the best dose of pazopanib hydrochloride in treating patients with solid tumors that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) or does not respond to treatment (refractory). Pazopanib hydrochloride may prevent the growth of new blood vessels that tumors need to grow. Studying samples of blood in the laboratory from patients receiving pazopanib hydrochloride may help doctors learn more about the effects of the body on the drug. It may also help doctors understand how well patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility and safety of individualizing pazopanib (pazopanib hydrochloride) monotherapy based upon attained pazopanib plasma concentrations so as to achieve desired target pazopanib plasma concentration in the highest possible fraction of treated patients.

SECONDARY OBJECTIVES:

I. To assess whether patient cytochrome P450 (CYP) or other polymorphisms may correlate with attained pazopanib levels in response to standard pazopanib dosing.

II. To assess whether patient trough pazopanib levels attained 24 hours after initiation of 800 mg daily fasting may predict steady state trough pazopanib levels after 14 days of pazopanib administration.

III. To assess whether patient trough pazopanib levels may correlate with observed pazopanib toxicities.

OUTLINE: This is a dose-escalation study.

Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Course length can be extended to 56 days at the discretion of the treating physician after 12 courses (1 year) of treatment on study.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of cancer which is now not amenable to alternative curative or clearly superior standard treatment options
* Measurable disease
* Hemoglobin (Hgb) >= 8.0 g/dL
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelet (PLT) = 100,000/uL
* Activated partial thromboplastin time (APTT) < 1.2 times upper limit of normal (ULN); (Note: use of warfarin is prohibited; low molecular weight heparin is allowed, so long as these criteria are met)
* International normalized ratio (INR) < 1.2 times ULN; (Note: use of warfarin is prohibited; low molecular weight heparin is allowed, so long as these criteria are met)
* Direct bilirubin =< 1.5 X upper limit of normal (ULN) (subjects with Gilbert's syndrome and elevations of indirect bilirubin only are eligible)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 X ULN
* Creatinine =< 1.5 times ULN OR measured creatinine clearance of >= 60 mL/min 1.73 m^2
* Urine protein/creatinine ratio < 1 or 24-hour urine < 1 gram
* < Grade 2 hypo/hyperkalemia
* < Grade 3 hypo/hypercalcemia
* < Grade 3 hypo/hyperphosphatemia
* < Grade 3 hypo/hypermagnesemia
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Ability to provide informed consent
* Willing to return to Mayo Clinic for follow up
* Life expectancy >= 84 days (3 months)
* Willingness to provide mandatory blood samples for pazopanib drug level assessments required for dosage adjustments, as well as for required pharmacogenomic studies
* Women of childbearing potential only: negative serum pregnancy test done =< 14 days prior to registration

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Corrected QT interval (QTc) >= 480 msec and/or receiving any concomitant medications that are associated with a risk of QTc prolongation and/or torsades de pointes; NOTE: these medications should be discontinued or replaced with drugs that do not carry these risks
* Subjects with any of the following cardiovascular conditions within the past 6 months

  * Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
  * Admission for unstable angina
  * Myocardial infarction
  * Cardiac angioplasty or stenting
  * Coronary artery bypass graft surgery
  * Pulmonary embolism, untreated deep venous thrombosis (DVT) or DVT which has been treated with therapeutic anticoagulation for less than 6 weeks
  * Arterial thrombosis
  * Symptomatic peripheral vascular disease
  * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; a subject who has a history of class II heart failure and is asymptomatic on treatment may be considered eligible
  * Active cardiac arrhythmia (except sinus arrhythmia, atrial fibrillation, asymptomatic premature ventricular contractions [PVCs])
  * Ejection fraction < institutional lower limit of normal (LLN) and/or history of cardiomyopathy
* Receiving a medication with known risk of torsades de pointes; the following medications are specifically prohibited: amiodarone, arsenic trioxide, bepridil, chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide, dofetilide, dolasetron, droperidol, erythromycin, halofantrine, haloperidol, ibutilide levomethadyl, mesoridazine, methadone, pentamidine, pimozide, procainamide, quinidine, sotalol, sparfloxacin, and thioridazine; patients should be watched carefully for indications of torsades de pointes, such as syncope; performing additional electrocardiograms (EKGs) on subjects who must take one or more of these medications is not required; however, additional investigations, including EKGs, may be performed as per the treating physician's judgment
* Blood pressure (BP) > 140 mmHg (systolic) and > 90 mmHg (diastolic); initiation or adjustment of BP medication is permitted prior to registration provided that the average of three BP readings at a visit prior to registration is < 140/90 mmHg
* Any of the following prior therapies:

  * Chemotherapy =< 28 days prior to registration
  * Mitomycin C/nitrosoureas =< 42 days prior to registration
  * Immunotherapy =< 28 days prior to registration
  * Biologic therapy =< 28 days prior to registration
  * Radiation therapy =< 28 days prior to registration
  * Radiation to > 25% of bone marrow
* Failure to fully recover from acute, reversible effects of prior chemotherapy (other anti-neoplastic therapy) and radiation therapy
* Subjects with known brain metastases
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation); Note: concomitant use of zoledronic acid, pamidronate or denosumab is allowed (and can be initiated while patients are on study therapy at investigator discretion)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive with cluster of differentiation (CD)4 counts < 200
* Receiving any other investigational agent
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history or prior malignancy, they must not be receiving other specific treatment (e.g. hormonal or chemotherapy) for their cancer
* Prior use of pazopanib (prior use of other kinase inhibitors allowed)
* Receiving any medications or substances that are strong or moderate inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) (indinavir, nelfinavir, atazanavir, ritonavir, clarithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, saquinavir, telithromycin, aprepitant, erythromycin, fluconazole, grapefruit juice, verapamil, diltiazem); use of the aforementioned strong or moderate inhibitors is prohibited < 7 days prior to registration
* Receiving any medications or substances that are inducers of CYP3A4 (efavirenz, nevirapine, carbamazepine, modafinil, phenobarbital, phenytoin, pioglitazone, rifabutin, rifampin, St. John's wort); use of the aforementioned inducers is prohibited =< 7 days prior to registration
* Receiving mitotane within 6 months of enrolling on the study
* Subjects with any condition that may impair the ability to swallow or absorb oral medications/investigational product including:

  * Any lesion, whether induced by tumor, radiation or other conditions, which makes it difficult to swallow capsules or pills
  * Prior surgical procedures affecting absorption including, but not limited to major resection of stomach or small bowel
  * Active peptic ulcer disease
  * Malabsorption syndrome
* Any of the following conditions:

  * Serious or non-healing wound, ulcer, or bone fracture
  * Current use of therapeutic warfarin; Note: low molecular weight heparin is allowed; prothrombin time (PT)/partial thromboplastin time (PTT) must meet the inclusion criteria
  * History of bleeding disorder, including patients afflicted with hemophilia, disseminated intravascular coagulation, or any other abnormality of coagulation potentially predisposing patients to bleeding
  * History of hemoptysis in excess of 2.5 mL (1/2 teaspoon ) within 8 weeks prior to first dose of study drug
  * Poorly controlled depression or anxiety disorder, or recent (=< 6 months) suicidal ideation
  * HIV-positive patients on combination antiretroviral therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Subjects with any condition that may increase the risk of gastrointestinal bleeding or gastrointestinal perforation, including

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesions
  * Inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or other gastrointestinal conditions which increase the risk of perforation
  * History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to beginning study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-03-19 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Biologically optimal dose (BOD) defined as the dose level and diet in combination that induces no toxicity requiring dose modification per protocol and achieves a satisfactory pazopanib trough concentration (Cmin greater than 30 ug/mL) | At 14 days
Adverse events profile, as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 3 months
  The number and severity of all adverse events (overall, by dose-level and diet, and by tumor group) will be tabulated and summarized.
Incidence of grade 3+ adverse events, as assessed by the NCI CTCAE version 4.0 | Up to 3 months
  The number and severity of grade 3+ adverse events will be tabulated and summarized.
Toxicity profile, as assessed by the NCI CTCAE version 4.0 | Up to 3 months
  Non-hematologic toxicities will be evaluated via the ordinal CTC standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Response profile, assessed using modified Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 3 months
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population The summary will be overall and by tumor group, and particularly by cohorts (first 34 patients vs. expansion cohort where a possibly refined definition of disease progression will be used).
Time until any treatment-related toxicity, as assessed by the NCI CTCAE version 4.0 | Up to 3 months
Time until treatment-related grade 3+ toxicity, as assessed by the NCI CTCAE version 4.0 | Up to 3 months
Time until hematologic nadirs (ANC, platelets, hemoglobin) , as assessed by the NCI CTCAE version 4.0 | Up to 3 months
Time to progression according to RECIST version 1.1 | Up to 3 months
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 3 months

SECONDARY OUTCOMES:
Pazopanib hydrochloride levels attained in response to standard dosing | At baseline, at 24 hours after pazopanib hydrochloride and day 14 of course 1, and at 14 days of dosage change
  Descriptive statistics, simple scatter plots and linear regression model will form the basis of presentation of these data. Attained levels will be correlated with cytochrome P450 and other polymorphisms and with observed toxicities.
Steady state pazopanib hydrochloride trough levels | 24 hours after initiation of 800 mg daily fasting
  Descriptive statistics, simple scatter plots and linear regression model will form the basis of presentation of these data. Will be correlated with steady state trough levels after 14 days.
Trough pazopanib hydrochloride levels | After 14 days of pazopanib hydrochloride administration
  Descriptive statistics, simple scatter plots and linear regression model will form the basis of presentation of these data. Trough levels will be correlated with observed toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Keith C Bible, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota